CLINICAL TRIAL: NCT04248504
Title: Digital Genetic Assistant (DGA) for Expanded Carrier Screening
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Igentify Ltd (Industry)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: MOH_2020-01-16_008638
Record Dates: First submitted 2020-01-16; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Genetic Disease
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Digital Genetic Assistant — An end-to-end digital solution to the carrier screening process from participant registration to receipt of the test results and their interpretations. These steps are provided using personalized animated videos.

SUMMARY:
The DGA provides an end-to-end digital solution to the preconception carrier screening process from participant registration to receipt of the test results and their interpretations. These steps are provided using personalized animated videos.

DETAILED DESCRIPTION:
Enrollment: The participant enrolls in the system prior to the visit and enters personal information into the DGA system. This step is estimated to takes approximately ten minutes and is expected to save valuable time should participants be required to come for a genetic counseling session. The medical questionnaire will self-adjust to address the clinical scenario related to each participant. This component will allow the attending physician to receive virtually all required information about the participant prior to their meeting, thereby improving communication with the participants, and potentially referring them to relevant tests even prior to their meeting. In the face-to-face meeting of the participants with the medical professional, most of the report summarizing treatment and family history, which the medical professional would have usually spent precious time filling, will be automatically ready, allowing for easy editing and finalization.

Next, the participant is guided through an on-line introductory personalized video explaining the genetic test and its implications tailored to the medical information that the participant entered in the questionnaire. The participant's understanding of the information presented in the personalized introductory video is tested by three questions. The participant must accurately answer the three questions. If the participant makes two mistakes the application opens the video in the relevant section and then asks the participant again. Following a successful completion of this step the participant is invited to sign an electronic Informed Consent to carry out the routine CarrierScan screening test (which is not a part of this study). The participants will re-sign a hard copy Informed Consent upon arrival to the Sheba Genetic Institute. A dedicated dashboard enables medical staff to monitor the progression of a participant along the process.

The Steps:

Step 1. Registration: During the initial phone call with potential participants, qualified staff that are part of the study will explain the process and extend an invitation to participated in the study. The DGA process will begin when the Sheba Medical Center (MC) Genetics Institute will send potential participants a link following the initial phone call between them. This link will enable the participant a secure connection to the DGA system. During the initial registration to the system the participant will undergo authentication using the standard two-factor authentication method based on phone number and the last four digits of the ID number of the participant. At the end of this process a new user will be created in the system.

Step 2. Interactive medical questionnaire: The interactive medical questionnaire is defined as the process of gathering personal information relevant to the specific clinical genetic scenario (e.g. personal information, personal and family medical information). The interactive medical questionnaire incorporated in the Enrollment app is based on Ministry of Health (MOH) guidelines for carrier screening. The questionnaire is dynamic and is interactively adapted based on live information supplied by the participant. In addition, the questionnaire is taking advantage of "natural language form", a user experience technique for drafting the questions, for a higher compliance rate. The questionnaire was approved by the Sheba MC PI.

Please note that the essence of the DGA system is to enable to conduct genetically relevant medical informatics processes in the context of digital sessions with secured and adaptive systems. Such data collection, pedigree drawing, and risk calculation takes place during face-to-face or over the phone meetings with medical staff using the currently practiced genetics counseling paradigm.

Step 3. Sample submission and signing a hard copy Informed Consent for the CarrierScan test: At the Sheba MC Genetic Institute, before the submission of buccal/saliva/blood samples to the test, participants will be asked to sign a hard copy Informed Consent.

Note: The CarrierScan screening test in not part of this study.

Step 4. Introductory personalized animated video: A personalized and dynamic animated video is machine-generated following a well-characterized medically supervised algorithm to tailor the video to each participant. The algorithm that generates the personalized introductory video is approved by the Sheba medical staff. Participants will receive a short-animated video summarizing the medical process they are going through. The content of these videos is dynamic and in full alignment with the Sheba MC requirements.

Following the dynamic video, the system will examine participants' understanding by a short interactive quiz that summarizes the relevant topics presented in the video. If the user answers wrong twice, he or she will be directed to the section in the video that provides the information to answer correctly. It is important for the usability study to test the responsiveness of the participant to sign the electronic Informed Consent following the personalized introductory video. The investigators believe that this video will provide a clear and, in most cases, more thorough explanation than the common face-to-face explanation.

e-Learning (general information on genetics and preconception): Provides education to the participant on basic genetic principles and concepts by a series of short dynamic videos making up an e-learning center.

On Board Dashboard for the Medical Staff:

A user-friendly dashboard will be accessible to relevant approved medical staff. It will include all the information gathered from the participant during the completion of the on-line registration and questionnaire process. Once the participant concludes the session of Participant Enrollment (Pre-Test), all his/her data are presented on the medical staff dashboard. A genetic counselor will be able to accept, reject, and/or revise the data. Next, the genetic counselor will send the participant a signed summary letter (PDF) via the DGA system, in a secured protocol (just as in the initial connection of the participant to the Sheba MC application). This letter will present the information entered into the system by the participant and invite him/her to perform the genetic test. Using the standard two-factor authentication method based on phone number and the last four digits of the participants' ID number, the participants will be able to view the report.

Counseling rationale - the logics of the DGA system (the "brain"):

This module processes participant information gathered during the participant enrollment process in combination with the results of the CarrierScan screening test. Residual risk is calculated automatically, and the system is ready to preset the medical staff with its suggestion on how to proceed. The Genetic Counseling Dashboard presents the supervising clinician with all relevant information for their approval or for further comments and edits. The results of the genetic tests are uploaded to the Sheba MC secured cloud. All processes described in this section also take place in the secure Sheba MC cloud.

Note: Only anonymization information of participants will be transferred to Igentify for analysis, assessment and improvement of the system.

DGA Algorithm: Next, the system utilizes its medically supervised genetic algorithm to decide on the outcome of the genetic counseling (high or low risk). The algorithm takes advantage of all relevant information in the system including the predictions of the residual risk. The outcomes of the system are either a digital report generator (see next section) or in the cases of couples that have been found to be at high risk, an invitation to a face-to-face genetic counseling session.

Genetic Counseling Dashboard (to medical staff in Sheba MC): Presents all the information gathered from the participant to the relevant medical staff, enabling decision-making regarding participant outcomes. The dashboard will enable the medical staff to approve or reject the suggestion of the DGA algorithm with regards to the participant's risk and the subsequent process. The system will raise flags in cases that action is needed and will support the subsequent face-to-face/telephone genetic counseling with reporting tools.

Interface for genetic results: Enables the DGA to incorporate genetic results from various genetic tests. In the current study, the DGA will work only with results of tests done at the Sheba MC genetic lab for the expanded carrier screening (CarrierScan and Fragile-X tests).

Counseling Summary Session:

Once the clinician approves the suggested decision of the DGA algorithm, this module is responsible to generate two types of outputs. Low risk participants (namely couples that were not found to be carriers of mutations in the same genes) are approved to receive an automated digital report (personalized video), while high risk participants are urged to schedule a face-to-face genetic counseling session. In high risk cases, the genetic counselor will have the digital information provided by the participants and the genetic test results, to make the counseling process more effective. The threshold of high/low risk assignment is determined by the head of the Sheba Genetic Institute.

Digital Genetic Counseling Report Generator: This component generates an animated, personalized dynamic video and a hard copy report (in PDF format) summarizing the genetic counseling provided to the participant online. Using the standard two-factor authentication method based on phone number and the last four digits of the participants' ID number, the participants will be able to view the personalized video and download the reports.

This module is responsible to coherently convey all personal and mandatory messages compatible with the guidelines of the Sheba Genetic Institute. The report is machine-generated and approved by medical personnel before its disclosure to the participant.

Having the DGA video available to the participants will allow them to review it repeatedly, until full understanding of the topic is achieved, as self-assessed by the participant. Each review will be recorded for medico-legal purposes.

• Support for In-Person Genetic Counseling: Face-to-face genetic counseling for high-risk participants will be aided by the system. The system dashboards will present the genetic counselor with a full report containing all gathered information to-date, which will be augmented with digital tools, such as pedigree editor and short self-explanatory animated videos aimed to facilitate an effective session.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to undergo expanded preconception carrier screening (CarrierScan Screening Test).
* Participants willing to use the DGA as part of their genetic screening.
* Participants willing to fill up questionnaires about their experience and understanding of the genetic counseling and share their clinical and DGA usage data with the study personnel.
* Fluent in Hebrew or English.
* Couples (Male + Female) that plan to have children together.
* Age above 18.

Exclusion Criteria:

* Individuals that undergo bone marrow transplantation.
* Participants refusing to participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Couples (Male + Female) that plan to have children together.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
The number of post-test face-to-face/telephone genetic counseling sessions | One year
  The investigators expect a significant reduction in the number of post-test face-to-face/telephone genetic counseling sessions. The current practice of expanded carrier screening provides a genetic counseling session to each couple who one of them is found to be a carrier of a genetic disease. Following the CarrierScan, expanded carrier screening test, ~60% of the couples are expected to be carriers of at least one disease. Using the DGA, the investigators expect that in the vast majority of cases (>95%), when low risk is identified, the couple will be informed by the DGA without requiring a face-to-face/telephone session. The investigators expect that some of the low risk couples that received digital report will still request further counseling. The investigators estimate this fraction to be 10-20% of the low risk participants.

CONTACTS AND LOCATIONS:
Overall Officials: Hagit Baris-Feldman, MD, Principal Investigator — Tel Avib Sourasky Medical Center

IPD SHARING:
Plan to Share IPD: No